CLINICAL TRIAL: NCT01027013
Title: A Phase II, Prospective, Randomized, Double-masked, Parallel Group, Multi-center Study Assessing the Safety and Efficacy of 2% Rebamipide (OPC-12759) Compared to Placebo for the Treatment of Keratoconjunctivitis Sicca (Dry Eye)
Brief Title: Safety and Efficacy Study of Rebamipide 2% Ophthalmic Suspension in Patients With Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACU-RED-203
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye Syndromes; Keratoconjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — rebamipide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rebamipide 2% ophthalmic suspension (Experimental)
  Interventions: Drug: rebamipide 2% ophthalmic suspension
- Placebo eye drops (Placebo Comparator)
  Interventions: Drug: placebo eye drops

INTERVENTIONS:
Drug: rebamipide 2% ophthalmic suspension — Instill one drop in each eye four times daily for 12 weeks.
  Arms: rebamipide 2% ophthalmic suspension
Drug: placebo eye drops — Instill one drop in each eye four times daily for 12 weeks.
  Arms: Placebo eye drops

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of rebamipide 2% suspension for the treatment of patients with dry-eye.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of dry eye as defined by the protocol

Exclusion Criteria:

* Ongoing ocular disease that may interfere with study parameters.
* Inability to stop using topical ophthalmic medications throughout the duration of the study
* Inability to stop the use of contact lenses for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Total fluorescein corneal staining score | 4 weeks
Primary ocular discomfort | 4 weeks

SECONDARY OUTCOMES:
Dry eye symptoms | 12 weeks
Ocular staining | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Boman, MD, PhD, Study Director — Kubota Vision Inc.
Locations (5):
- United States (5):
  - The Eye Care Group, P.C., Waterbury, Connecticut
  - Richard Eiferman, MD, Louisville, Kentucky
  - Central Maine Eye Care, Lewiston, Maine
  - Ora, Inc, Andover, Massachusetts
  - Total Eye Care, P.A., Memphis, Tennessee